CLINICAL TRIAL: NCT00842790
Title: Medical and Economical Impact of Predicting the Response to Anti-angiogenic Treatment in Metastatic Renal Cell Carcinoma Using Functional CT and MRI
Brief Title: Impact of Predicting Anti-angiogenic Response in mRCC Using Functional Imaging
Acronym: REMISCAN
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P060407
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2009-02

CONDITIONS: Carcinoma, Renal Cell
Keywords: Carcinoma, Renal Cell [C04.557.470.200.025.390]; Angiogenesis Inhibitors [D27.505.954.248.025]; Tomography Scanners, X-Ray Computed [E07.913]; Magnetic Resonance Imaging [E01.370.350.825.500]; Diffusion Magnetic Resonance Imaging [E01.370.350.825.500.150]; Perfusion [E05.680]
MeSH Terms: conditions — Carcinoma, Renal Cell; Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal is to study the impact of functional MRI and CT evaluation of changes in tumor vessels induced by anti-angiogenic treatment in patients with metastatic RCC.

The hypothesis is that good responders and poor responders will have different responses induced by anti-angiogenic treatment, and that the detection of theses changes by functional imaging can improve the therapeutic management.

Functional CT and MRI will be performed in 200 patients before the beginning of antiangiogenic treatment, 7 days after and every 6 week until tumor progression (as defined by the RECIST criteria). Perfusion and diffusion parameters will be measured using a dedicated software.

DETAILED DESCRIPTION:
The aim is to evaluate the capacity of functional CT and functional MRI to measure reliable biomarkers capable of evaluating the efficacy of anti-angiogenic treatment.

Patient and methods

- Patients 200 patients with metastatic RCC will be enrolled in the study. Patients will be recruited by an oncologist and the images will be acquired by a radiologist.

Patients will be followed until tumor progression (as defined by RECIST) or during 2 years following inclusion if there is no progression.

- Imaging data acquisition Morphological and functional imaging will be obtained before the beginning of the anti-angiogenic treatment, at 7±2 days and every 6 weeks until tumor progression.

Progression is defined following the RECIST criteria.

* CT examination will be have two parts: the first one will be a dynamic acquisition during 3 min (using low kV)focused on a "functional target lesion" during bolus injection of a contrast agent for functional analysis, and the second one will be a morphologic acquisition over the chest, the abdomen and the pelvis for RECIST evaluation.
* MRI examination will have two parts: the first one will be a diffusion weighted sequence focused on the same functional target as the one imaged on CT, and the second one will be a dynamic acquisition using a T1 weighted gradient echo sequence with less than 4 s sampling time during 5min following the bolus injection of contrast agent.

  * Imaging data analysis The examinations will be anonymized and transferred to a workstation for processing. Images will be processed by two independent readers.

Diffusion coefficient maps will be obtained using linear regression. The microvascular parametric maps yielding as tissue blood flow, tissue blood volume, mean transit time, permeability surface area product and tissue interstitial volume will be calculated for both the CT and MRI dynamic series using a proprietary software by means of compartmental modeling with an arterial input function (AIF).

Mean parameters will be recorded for different regions of interest (ROI) in the tumors (whole tumor, periphery, center).

Morphological CT images will be analyzed following the RECIST criteria.

-Statistical analysis The functional parameters will be analyzed for inter-observer reproducibility. The correlation between parameters obtained using functional CT and functional MRI will tested.

Patients will be classified as good responders and poor responders according to RECIST follow-up.

The correlation between each baseline functional parameter and the RECIST response will be tested to evaluate the usefulness of the baseline parameters as predictors of response.

The correlation between each parameter's changes under treatment as compared to the baseline value will be tested to evaluate the efficacy of each parameter to detect the response to the anti-angiogenic drug. The precocity of the detection of the response using the parameter variations will be also tested.

Finally, the economical impact of the use of the microvascular parameters as biomarkers of treatment efficacy will be tested.

ELIGIBILITY:
Inclusion Criteria:

* with metastatic RCC
* without previous recent antiangiogenic treatment

Exclusion Criteria:

* severe renal insufficiency
* allergy to contrast agents
* pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: oncologic hospital visit
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2008-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
RECIST criteria evolution | at day 7 and after every 6 at 16 weeks during 2 years
  time-to-progression with anti-angiogenic traitment evaluated by RECIST criteria

SECONDARY OUTCOMES:
Validation of the technical and acquisition measurement models | at day 7 and after every 6 at 16 weeks during 2 years
  Validation of the technical and acquisition measurement models of tumor perfusion MRI and CT, and diffusion MRI, study of reproducibility
Assessment of potential drug costs | at the end
  Assessment of potential drug costs avoided by use of innovative prognostic criteria for adapting treatment

CONTACTS AND LOCATIONS:
Overall Officials: Stephane OUDARD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris; Charles-André Cuenod, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- service of oncology- HEGP, Paris, France